CLINICAL TRIAL: NCT05193812
Title: Predicitve Value of Copeptin In CO-intoxicated Patients
Brief Title: Predicitve Value of Copeptin In CO-intoxicated Patients - A Prospective Cohort Study
Acronym: ALCOPOP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1726
Record Dates: First submitted 2021-11-26; First posted 2022-01-18 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: CO Poisoning
Keywords: carbon monoxide; intoxication; disability-free survival
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ALCOPOP is a prospective cohort study entitled "Predicitve Value of Copeptin in CO-intoxicated Patients". The primary objective of this study is to assess the independent association between early Copeptin and / or Troponin concentrations at presentation at the emergency department with disability-free survival after carbon monoxide (CO) -intoxication. Further secondary aims are to determine the independent association between early postoperative Copeptin and / or Troponin concentrations and major adverse cardiovascular events (MACE), mortality and long-term neurological outcome.

Adult patients with acute CO-intoxication (CO-hemoglobin >10%) will be included. Main exposure will be Copeptin and Troponin concentrations. Primary endpoint will be disability-free survival at 90 days. The investigators assume to include 120 patients in 24 months

DETAILED DESCRIPTION:
Aims of the study

To evaluate early Copeptin at arrival at emergency department based on the following:

1. Discrimination for 90-day-disability-free survival (primary), 30-day-disability-free survival (secondary) and for 30-day and 90-day MACE, 30-day and 90-day all-cause mortality (secondary) as well as 30-day and 90-day-neurological outcome (secondary) and length of hospital stay (secondary).
2. Independent association with 90-day disability-free survival (primary), days alive out of hospital at 30 days and 90 days (secondary) and MACE at 30 days and 90 days after CO-intoxication, 30-day and 90-day all-cause mortality and (secondary) as well as the 30-day and 90-day neurological outcome (secondary) and length of hospital stay (secondary).

To evaluate early Troponin at arrival at emergency department in terms of:

1. Discrimination for 90-day disability-free survival (primary), 30-day-disability-free survival (second) and for 30-day and 90-day MACE as well as 30-day and 90-day all- cause mortality (secondary) and length of hospital stay (secondary).
2. Independent association with 90-day-disability-free survival (primary), days alive out of hospital at 30 days and 90 days (secondary) and MACE at 30 days and 90 days after CO-intoxication as well as 30-day and 90 days all-cause mortality (secondary) and length of hospital stay (secondary).

The initial patient visit will take place after screening of patients and eligibility assessment and no later than on the day after admission to the emergency department (day +1). After provision of patient information and written informed consent, baseline data will be extracted from clinical source documents. The investigators plan to sample blood upon arrival in the emergency department (Troponin and Copeptin), and on day 1 and 2 after CO-intoxication (Troponin). Another blood sample will be carried out after hyperbaric oxygen (HBO) therapy to obtain a a second Copeptin measurement. Sampling will occur as far as possible concurrently to clinically indicated blood samples. Blood samples will be analyzed in a certified laboratory.

The investigators will contact all patients after 30 days and 90 days by postal mail and/or phone call (personnel blinded to biomarkers concentrations) to obtain for the 12-item WHO Disability Assessment Schedule (WHODAS) 2.0 and information on potential events. In case of the report of potential endpoints, the patient's general practitioner and/or treating hospital will be contacted for more detailed information and source documents for MACE, persistent neurological sequelae (PNS) and delayed neurological sequela (DNS) adjudication. Adjudicators will be trained in the study definitions and blinded to biomarkers concentrations.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with acute CO-poisoning, defined as CO-Hb levels >10%

Exclusion Criteria:

* Unwilling or unable to provide consent
* Inability to follow the procedures of the study, e.g. due to language barriers, psychiatric disorders, dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The University Hospital Duesseldorf is one of three centres for hyperbaric oxygen therapy (HBO) in western Germany treating about 60-100 patients with CO-intoxication annually. we will screen each patient with CO-intoxication admitted to the emergency department of the Univerisity Hospital Duesseldorf.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
disability-free survival | 90 days
  Disability is defined as a persistent impairment in health status, as measured by the 12-item WHO Disability Assessment Schedule (WHODAS) 2.0 score, of at least 24 points when using response scores of 1-5 for each item, reflecting a disability level of at least 25% and being the threshold point between 'disabled' and 'not disabled' as per WHO guideline.

SECONDARY OUTCOMES:
Disability-free survival at 30 days after CO-intoxication | 30 days
  Disability is defined as a persistent (at least 1 month) impairment in health status, as measured by the 12-item WHODAS 2.0 score, of at least 24 points when using response scores of 1-5 for each item, reflecting a disability level of at least 25% and being the threshold point between 'disabled' and 'not disabled' as per WHO guideline.
WHODAS 2.0 Score at 30 and 90 days after CO-intoxication | 30 and 90 days
  12-item WHODAS 2.0 score
Days alive and out of hospital at 30 days and 90 days after CO-intoxication | 30 and 90 days
  patient centred outcome; amount of days spent at home after CO-intoxication
MACE at 30 days and 90 days | 30 and 90 days
  defined as non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure or transfer to a higher unit of care, atrial fibrillation or stroke
All-cause mortality at 30 days and 90 days | 30 and 90 days
  mortality after CO-intoxication independent of its cause
Length of hospital stay | from admission (day informed consent was given) until day of hospital discharge of the respective participant, up to 90 days
  amount of days spent at hospital
Length of ICU-stay | from admission (day informed consent was given) until day of hospital discharge of the respective participant, up to 90 days
  amount of days spent at ICU
Persistent neurological sequelae (PNS) at 30 days and 90 days measured by a questionnaire | 30 days and 90 days
  Symptoms or signs attributable to CO poisoning that are evident immediately following poisoning including subtle personality changes, mood disorders headaches, tiredness, difficulty in concentrating, difficulty in sleeping, visual disorders, and new difficulties with social or professional activities and memory impairment to (much less commonly) focal neurological injuries and other severely disabling manifestations of hypoxic brain injury
Delayed neurological sequelae (DNS) at 30 days and 90 days measured by a questionnaire | 30 days and 90 days
  Symptoms and signs as mentioned above (see outcome 9) occurring between hospital discharge and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: PD Stephan Sixt, Principal Investigator — Department of Anaesthesiology, University Hospital Duesseldorf